CLINICAL TRIAL: NCT02664649
Title: Anti-Thrombotic Strategy to Lower All Cardiovascular and Neurologic Ischemic and Hemorrhagic Events After Trans-Aortic Valve Implantation for Aortic Stenosis
Brief Title: Anti-Thrombotic Strategy After Trans-Aortic Valve Implantation for Aortic Stenosis
Acronym: ATLANTIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Action Research Group (Other); Bristol-Meyers Squibb & Pfizer (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P141102; 2015-001676-21 (EudraCT Number)
Record Dates: First submitted 2015-09-30; First posted 2016-01-27 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Symptomatic Aortic Stenosis; Eligible for Transcatheter Aortic Valve Replacement
Keywords: TAVR; Apixaban; Anticoagulant; VKA; Antiplatelet therapy; Aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — apixaban; Factor Xa Inhibitors; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apixaban (Experimental): Investigational Product is open label apixaban 5 mg tablets taken orally two times a day for 12 months. Subjects with 2 or more of the following characteristics will take apixaban 2.5 mg tablets orally twice daily: age ≥80 years, body weight <60 kg, serum creatinine ≥1.5 mg/dL [133 μMol/L].
  - Also, subjects with severe renal insufficiency [calculated Creatinine Clearance (Cr.Cl.) (Cockroft-Gault) between 15-29 ml/min] will take apixaban 2.5 mg tablets orally twice daily
  Interventions: Drug: Apixaban
- Standard of care (Active Comparator): VKA or Antiplatelet therapy
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Apixaban — Investigational Product is open label apixaban 5 mg tablets taken orally two times a day for 12 months. Subjects with 2 or more of the following characteristics will take apixaban 2.5 mg tablets orally twice daily: age ≥80 years, body weight <60 kg, serum creatinine ≥1.5 mg/dL [133 μMol/L].
  - Also, subjects with severe renal insufficiency [calculated Creatinine Clearance (Cr.Cl.) (Cockroft-Gault) between 15-29 ml/min] will take apixaban 2.5 mg tablets orally twice daily
  Other Names: Brand name : Eliquis drug class : anticoagulant, factor-Xa inhibitor
  Arms: Apixaban
Drug: Standard of care — VKA or Antiplatelet therapy
  Arms: Standard of care

SUMMARY:
ATLANTIS is a multicenter, phase IIIb, prospective, open-label, randomized trial.

The objective of this study is to demonstrate superiority of a strategy of anticoagulation with apixaban (Anti-Xa Group) as compared to the current standard of care in patients who have undergone a successful TAVI procedure.

The randomization is stratified according to the presence or not of a mandatory indication for anticoagulation for a reason other than the TAVI procedure (e.g. atrial fibrillation or DVT/PE).

DETAILED DESCRIPTION:
Guidelines on antithrombotic therapy after TAVI are scarce and no randomized evaluation has been performed to demonstrate what the optimal antithrombotic strategy is. The rates of major stroke and of major bleeding on DAPT, the standard of care in TAVI (Class IIb LOE C), are respectively as high as 3% and 10% within the first 30 days excluding the perioperative period. In addition, the rate of MACCE is estimated to be of 15% on DAPT. However, more than half of senior patients display high on-clopidogrel platelet reactivity, less than 1/3 undergo coronary stent implantation prior to valve replacement and more than 1/3 display transient atrial fibrillation (AF) during hospital stay. Anticoagulation appears therefore to be underused in this high stroke risk population and has never been evaluated in post-TAVI procedures. Non-vitamin K Oral Anticoagulants (NOAC) have shown superiority or non-inferiority versus VKA to prevent cardio-embolic events with a consistent reduction in intracranial bleeds in patients with non-valvular AF. Apixaban, a direct anti-Xa inhibitor, is the only NOAC which has demonstrated a mortality benefit associated with significant reductions in embolism and major bleeding versus VKA. In addition, apixaban is the only NOAC which has demonstrated superiority over aspirin to prevent cardio-embolic events with a similar safety profile in non-valvular AF patients with a contraindication to VKA. The investigators therefore formulate the hypothesis that apixaban is superior to SOC to prevent cardiovascular events in post-TAVI procedures.

The main purpose is to demonstrate superiority of a strategy of anticoagulation with apixaban 5mg bid (Anti-Xa Group) with dose adjustment as compared to the current standard of care (SOC Group = VKA or Antiplatelet therapy) as measured by the time from randomization to the first occurrence of any event of the composite endpoint of death, myocardial infarction, stroke/TIA/systemic embolism, intracardiac or bioprosthesis thrombus, episode of deep vein thrombosis or pulmonary embolism, life-threatening or disabling or major bleeding at one year follow-up defined according to VARC2.

Patients who underwent a clinically successful TAVI procedure. Non-inclusion criteria include any recent acute cardiovascular event, mechanical heart valve, necessary use of prasugrel or ticagrelor (new P2Y12 inhibitors), concomitant medical illness associated with reduced survival, end stage renal failure defined as a creatinine clearance < 15mL/min.

ELIGIBILITY:
Inclusion Criteria:

* All patients after clinically successful TAVI procedures irrespective of prior antithrombotic treatment are eligible for randomization.
* Ability to understand and to comply with the study protocol.
* Written informed consent.
* Men and women ≥18 years of age.

Non-inclusion Criteria:

* Creatinine Clearance < 15mL/min (Cockcroft formula) or patient undergoing dialysis.
* Mechanical valves.
* Known severe mitral valve stenosis requiring an intervention.
* Unsuccessful TAVI requiring re-intervention.
* Ongoing major bleeding or vascular complication (patients may become candidate to the study once stabilized).
* Prior history of intracranial haemorrhage.
* Recent cerebro-vascular event (CVE) or transient ischemic attack on anticoagulant therapy (<6 weeks).
* Cardiogenic shock manifested by low cardiac output, vasopressor or respiratory dependence, or mechanical hemodynamic support.
* Planned major surgery during follow-up defined as high-bleeding risk according to ESC/EHRA and requiring interruption of the study drug with bridging
* Concomitant medical illness (terminal malignancy) that is associated with expected survival less than one year.
* Concomitant use of prasugrel or ticagrelor.
* Following concomitant treatments that are potent inhibitors of CYP3A4: azole antifungals (itracozanole and ketoconazole), macrolide antibiotics (clarithromycine and telithromycin), and protease inhibitors (ritonavir, indinavir, nelfinavir and aquinavir) and nefazadone.
* Women of childbearing potential (WOCBP)*.
* Men who are sexually active with WOCBP* partners.

  *Any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over age 45 in the absence of other biological or physiological causes
* Pregnancy and breast feeding.
* Currently participating in an investigational drug or another device trial within the previous 30 days.
* Known Liver affection associated with coagulopathy and medical significant risk of bleeding.
* Uncontrolled cancer with life expectancy of less than one year.
* Inability to give informed consent or high likelihood of being unavailable for follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1510 (Estimated)
Dates: Start 2016-08-26 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Composite of death, myocardial infarction, stroke, systemic embolism, intracardiac or bioprosthesis thrombus, any episode of deep vein thrombosis or pulmonary embolism, life-threatening or disabling or major bleeding at one year follow-up. | up to 13 months
  life-threatening or disabling or major bleeding defined according to VARC-2 definitions over one year follow-up.

SECONDARY OUTCOMES:
Presence or not of an indication (other than TAVI) for anticoagulation described in the medical record. | from screening to randomization
  Information present in the medical record of the patient
First occurrence of any event of the following composite criteria: a) Death, MI, any stroke through one year of randomization, b) Death, any stroke/TIA or systemic embolism c) Each individual parameter of the primary endpoint | up to 13 months
  life-threatening (including fatal) or disabling or major bleeding (BARC 4, 3a, b and c) (primary safety endpoint) as defined according to VARC-2.
Minor bleedings (BARC 2 or 3a) | up to 13 months
  occurrence of any Minor bleedings (BARC 2 or 3a)
Any bleeding | up to 13 months
  occurrence of any bleeding
Any evidence for valve thrombosis including hypoattenuated leaflet thickening (HALT) | up to 13 months
  Valve thrombosis including hypoattenuated leaflet thickening (according to ETT results)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe COLLET, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (4):
- ACTION Study Group, Institut de Cardiologie, Centre Hospitalier Universitaire Pitié Salpêtrière (APHP), UPMC, Paris, France
- Division of Cardiology and Angiology II, University Heart Center Freiburg, Bad Krozingen, Südring 15, Germany
- Unità Operativa di Cardiologia Fondazione Gabriele Monasterio C.N.R., Massa, Via Aurelia Sud, Italy
- Hospitalet de Llobregat-Hospital Universitari de Bellvitge, Barcelona, Cardiologia Feixa Llarga, S/n, Spain

REFERENCES:
- [Derived] Montalescot G, Redheuil A, Vincent F, Desch S, De Benedictis M, Eltchaninoff H, Trenk D, Serfaty JM, Charpentier E, Bouazizi K, Prigent M, Guedeney P, Salloum T, Berti S, Cequier A, Lefevre T, Leprince P, Silvain J, Van Belle E, Neumann FJ, Portal JJ, Vicaut E, Collet JP; ATLANTIS Investigators of the ACTION Group. Apixaban and Valve Thrombosis After Transcatheter Aortic Valve Replacement: The ATLANTIS-4D-CT Randomized Clinical Trial Substudy. JACC Cardiovasc Interv. 2022 Sep 26;15(18):1794-1804. doi: 10.1016/j.jcin.2022.07.014. Epub 2022 Aug 31. PMID 36137682
- [Derived] Collet JP, Van Belle E, Thiele H, Berti S, Lhermusier T, Manigold T, Neumann FJ, Gilard M, Attias D, Beygui F, Cequier A, Alfonso F, Aubry P, Baronnet F, Ederhy S, Kasty ME, Kerneis M, Barthelemy O, Lefevre T, Leprince P, Redheuil A, Henry P, Portal JJ, Vicaut E, Montalescot G; ATLANTIS Investigators of the ACTION Group. Apixaban vs. standard of care after transcatheter aortic valve implantation: the ATLANTIS trial. Eur Heart J. 2022 Aug 1;43(29):2783-2797. doi: 10.1093/eurheartj/ehac242. PMID 35583186
- [Derived] Collet JP, Berti S, Cequier A, Van Belle E, Lefevre T, Leprince P, Neumann FJ, Vicaut E, Montalescot G. Oral anti-Xa anticoagulation after trans-aortic valve implantation for aortic stenosis: The randomized ATLANTIS trial. Am Heart J. 2018 Jun;200:44-50. doi: 10.1016/j.ahj.2018.03.008. Epub 2018 Mar 10. PMID 29898848
- [Derived] Piayda K, Zeus T, Sievert H, Kelm M, Polzin A. Subclinical leaflet thrombosis. Lancet. 2018 Mar 10;391(10124):937-938. doi: 10.1016/S0140-6736(18)30534-8. No abstract available. PMID 29536857